CLINICAL TRIAL: NCT07272356
Title: Investigation of the Efficacy of Local Minimally Invasive Ablative Therapy for Pulmonary Tumors and Its Impact on Respiratory Function
Brief Title: Evaluation of Efficacy of Minimally Invasive Local Therapy for Lung Tumors and Its Impact on Breathing Function
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aurimas Macionis (Other)
Responsible Party: Sponsor-Investigator, Aurimas Macionis, Principal Investigator, Lithuanian University of Health Sciences
Organization: Lithuanian University of Health Sciences (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-BE-10-0015
Record Dates: First submitted 2025-09-28; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer (Non-Small Cell); Lung Metastases From Any Primary
Keywords: non-small cell lung cancer; lung metastases; image-guided thermal ablation; surgery; microwave ablation; cryoablation; stereotactic body radiotherapy; cancer recurrence; quality-of-life; oncologic control; respiratory function
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Respiratory Aspiration | interventions — Surgical Procedures, Operative; Anterior Temporal Lobectomy; Cryosurgery; Radiosurgery; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Surgery (Active Comparator): Surgical treatment with the aim of complete tumor removal with safety margins. The procedures may include lobectomies, segmentectomies, atypical resections, or pneumonectomies. The surgery may or may not include regional lymph node dissection.
  Interventions: Procedure: Surgery
- SBRT (Active Comparator): Stereotactic body radiation therapy (SBRT) will be performed with the aim of radical tumor eradication by delivering very high doses of radiation to the tumor. Dose and fractionation regimens will be individualized, with a target median BED₁₀ of 100 Gy.
  Interventions: Radiation: SBRT
- Ablation (Active Comparator): Image-guided thermal ablation is a minimally invasive treatment aiming for radical tumor destruction using either heat or cold. In this trial, procedures include microwave ablation and cryoablation, all performed under general anaesthesia with CT guidance to ensure complete lesion coverage and adequate safety margins.
  Interventions: Procedure: Ablation

INTERVENTIONS:
Procedure: Surgery — Surgical resection performed under general anaesthesia, including lobectomy, segmentectomy, or atypical resection. All anatomical resections were accompanied by lymph node dissection, while atypical resections were performed without lymph node removal. Procedures were carried out via open thoracotomy, with some performed through mini-thoracotomy.
  Other Names: Lobectomy; Anatomical resection; Atypical resection; Segmentenctomy
  Arms: Surgery
Procedure: Ablation — Image-guided thermal ablation performed under general anaesthesia with CT guidance, including microwave ablation (TATO2 system, single or overlapping insertions) and cryoablation (CryoCare Touch™ system, three freeze-thaw cycles). Tract sealing was performed to minimize complications.
  Other Names: Microwave ablation; Cryoablation
  Arms: Ablation
Radiation: SBRT — Stereotactic body radiation therapy delivered with a Varian TrueBeam™ linear accelerator, using 4D-CT planning, daily cone-beam CT image guidance, RTOG-based organ-at-risk constraints, and individualized fractionation regimens with the aim of a median biologically effective dose of 100 Gy.
  Other Names: Stereotactic body radiotherapy; Radiotherapy
  Arms: SBRT

SUMMARY:
This clinical study is evaluating different treatment options for patients with malignant lung tumors, including both primary lung cancer and tumors that have spread to the lungs from other parts of the body. The goal is to compare the safety, effectiveness, and quality-of-life impact of three approaches: surgery, stereotactic body radiotherapy (SBRT), and minimally invasive thermal ablation (microwave or cryoablation).

Thermal ablation is a procedure in which a small antenna is inserted through the skin into the tumor and the cancer cells are destroyed using heat or freezing. SBRT uses precisely targeted radiation to destroy tumors, while surgery involves removing part of the lung. These methods are already used in routine care, but this study directly compares them to understand which patients may benefit most from each approach.

In addition to cancer control, the study is measuring how these treatments affect breathing function. Patients will have regular follow-up visits with CT scans, breathing tests, and blood draws for up to two years.

About 100 adults in Lithuania are expected to participate. The results will help doctors make better treatment recommendations, balancing cancer control with patient well-being, lung function, and quality of life.

DETAILED DESCRIPTION:
Lung cancer remains one of the leading causes of cancer-related death worldwide, and the lungs are also a common site of metastases from other cancers such as colorectal, breast, or kidney tumors. While surgery is considered the gold standard for treatment of early-stage lung cancer and resectable pulmonary metastases, many patients are not suitable surgical candidates due to age, comorbidities, or personal choice. For these patients, less invasive treatments such as stereotactic body radiotherapy (SBRT) or image-guided thermal ablation may provide effective alternatives.

This study is designed to evaluate the safety, effectiveness, and patient-centered outcomes of three treatment strategies for malignant lung tumors:

* Surgery (anatomical lung resection, when feasible)
* Stereotactic body radiotherapy (SBRT), which delivers high doses of precisely targeted radiation
* Minimally invasive thermal ablation, performed under CT guidance using microwave or cryoablation technology to destroy tumor tissue with heat or freezing

Thermal ablation and SBRT are established treatment options in many centers worldwide, but there is limited prospective data directly comparing these modalities with surgery. This trial aims to address that gap by examining not only oncologic outcomes such as recurrence, survival, and complications, but also functional and quality-of-life outcomes.

Study Objectives:

* To compare disease control (local, regional, and distant recurrence) and survival outcomes across surgery, SBRT, and ablation.
* To evaluate complication rates and hospitalization needs after each treatment.
* To assess the effect of each treatment on respiratory function using spirometry, gas diffusion testing, and lung perfusion scintigraphy.
* To monitor health-related quality of life (HRQoL) using the SF-36 questionnaire before and after treatment.

Study Design:

This is a prospective, single-center, non-randomized study conducted at the Lithuanian University of Health Sciences Kaunas Clinics. Eligible patients are adults (≥18 years) with either primary peripheral lung cancer or oligometastatic pulmonary disease (≤5 lesions, each ≤3 cm in size), who are suitable for surgery, SBRT, or thermal ablation based on multidisciplinary team (MDT) assessment. Patients are assigned to one of the three treatment groups-surgery, SBRT, or ablation-based on clinical suitability and shared decision-making between the MDT and the patient.

Follow-Up Procedures:

Participants are followed for up to 24 months with scheduled visits and investigations, including:

* Clinical assessments at baseline, 1, 3, 6, 12, 18, and 24 months
* Chest CT scans at baseline and 1, 3, 6, 12, 18, and 24 months after the treatment
* FDG-PET/CT if clinically indicated
* Spirometry and gas diffusion testing at baseline, 3 months, and 6 months
* Lung perfusion scintigraphy at baseline and 3 months
* Blood sampling (up to 10 ml) at baseline, 3 months, and 6 months
* Completion of quality-of-life questionnaires at baseline and one month after treatment

Risks and Benefits:

Risks include discomfort from diagnostic procedures (blood draws, imaging, spirometry), possible treatment-related complications such as pneumothorax after ablation, infection or post-operative pain after surgery, and radiation-related side effects (e.g., radiation pneumonitis, infection) after SBRT. However, all procedures are well-established in clinical practice, and serious complications are rare. Benefits include close monitoring of disease status with imaging, which may enable early detection of recurrence and timely treatment. Patients may also benefit from comprehensive functional assessments that can guide future care.

Expected Outcomes:

This study is expected to provide comparative information on the safety, effectiveness, and impact on quality of life of surgery, stereotactic body radiotherapy, and minimally invasive thermal ablation in patients with malignant lung tumors. By evaluating recurrence, survival, complications, and respiratory function, the study aims to identify which patients benefit most from each treatment approach and to support more personalized treatment planning in the future.

Sample Size and Duration:

The study aims to enroll approximately 100 participants in Lithuania. Each participant will be followed for two years after treatment.

Significance:

This study is expected to provide valuable evidence on the comparative effectiveness of surgery, SBRT, and thermal ablation in the management of malignant pulmonary tumors. By integrating oncologic, functional, and quality-of-life outcomes, the study seeks to support personalized medicine approaches and improve decision-making in multidisciplinary care of lung cancer and metastases.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older)
* Verified systemic therapy-naive biopsy-proven NSCLC, stages from Tis to T2; or oligometastatic peripheral (≤ 5 lesions) lung disease;
* All lesions are ≤3 cm in size and accessible for surgery, ablation or SBRT;
* No local nodal or distant metastatic disease on diagnostic imaging;
* Documented agreement on the recommended curative treatment by a multidisciplinary team, including a pulmonologist, interventional radiologist, radiation therapist, thoracic surgeon, and oncologist;
* Documented patient's agreement to receive the intended therapy and to participate in this study via a signed informed consent form.

Exclusion Criteria:

* Central lung tumors (<2 cm from the main bronchi or hilum);
* >5 or diffuse lung lesions, or prior local treatment to the same lesion;
* Major comorbidities, physical or social limitations precluding trial participation;
* Contraindications to general anesthesia, inability to temporarily withdraw antiplatelet therapy, or evidence of severe coagulopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2026-06-14 (Estimated); Study Completion 2026-06-14 (Estimated)

PRIMARY OUTCOMES:
Local oncologic control | Up to 24 months after treatment.
  Evaluate and compare local relapse rates on CT or PET/CT imaging following surgery, stereotactic body radiotherapy (SBRT), or thermal ablation. Local disease control is the central measure of treatment effectiveness.

SECONDARY OUTCOMES:
Disease Recurrence | Up to 24 months after treatment.
  Evaluate and compare regional and distant recurrence rates following surgery, stereotactic body radiotherapy (SBRT), or thermal ablation.
Survival | Up to 24 months after treatment
  Evaluate and compare disease-free survival (DFS) and overall survival (OS) following surgery, stereotactic body radiotherapy (SBRT), or thermal ablation.
Complication Rates | Immediately post-treatment and throughout the 24-month follow-up.
  Frequency, severity, and type of treatment-related complications, classified according to CIRSE (Cardiovascular and Interventional Radiological Society of Europe) standards.
Hospitalization | From the date of treatment until the date of discharge, assessed up to 24 months
  Length of hospital stay required for each treatment modality.
Respiratory Function: spirometry | Baseline before treatment and 3-12 months post-treatment.
  Changes in forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), and FEV1/FVC due to treatment. The values are described as absolute values (litres), percentages of predicted values, and z-scores.
Respiratory Function: gas diffusion | Baseline before treatment and 3-12 months post-treatment.
  Changes in forced expiratory volume in diffusing capacity of the lung for carbon monoxide, corrected for hemoglobin (DLCOc ) due to treatment. The values are described as mmol/min/kPa or % pred
Respiratory Function: lung perfusion scintigraphy | Baseline before treatment and 3-12 months post-treatment.
  Changes in lung lobar perfusion percentages on SPECT/CT due to treatment. Lobar perfusion percentages calculated from SPECT counts (total counts in a lobe / total counts in both lungs x 100), the data expressed in millilitres (mL).
Health-Related Quality of Life | At baseline and one month post-treatment.
  Changes in patient-reported outcomes using the 36-Item Short Form Health Survey (SF-36 questionnaire), focusing on physical, social, emotional, and mental health domains. The data of each domain is expressed in a score from 0 to 100, with 0 representing the poorest health status and 100 indicating the best possible health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian University of Health Sciences Kaunas Clinics, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Yes
Yes, de-identified IPD will be shared. IPD Types: Baseline demographics, tumor characteristics, treatment details, and outcome measures (local control, survival, toxicity).
  Supporting Documents: Study protocol, informed consent form.
Supporting Information: Study Protocol, ICF
Time Frame: Available starting 12 months after publication, and accessible for 3 years.
Access Criteria: Researchers with a methodologically sound proposal; requests to be submitted to Kaunas Regional Biomedical Research Ethics Committee:
  Lithuanian University of Health Sciences, Mickevičiaus g. 9, LT-44307, Kaunas Phone: +370 37 326889 Email: kaunorbtek@lsmuni.lt